CLINICAL TRIAL: NCT02291107
Title: Robot-assisted Gait Training in Patients Affected by Multiple Sclerosis: Rehabilitative Efficacy Evaluation and Comparison With Traditional Methods
Brief Title: Robot-assisted Gait Training in Patients With Multiple Sclerosis: Efficacy and Comparison With Traditional Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Habilita, Ospedale di Sarnico (Other)
Responsible Party: Principal Investigator, Dr. Cristiano Sconza, MD, Habilita, Ospedale di Sarnico
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LK.S P07
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis
Keywords: Gait orthosis; Lokomat; Robotic Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Participants received 25 sessions of robotically driven gait orthosis training on the Lokomat. Training occurred approximately 5 days/ week for 5 weeks, and each training session on the Lokomat lasted 30 minutes. All sessions were supervised by a trained research therapist. All participants started with 40% body weight-support and an initial treadmill speed of 1.5 km/h. Body weight-support was used primarily to facilitate an increase in walking speed; therefore, progression of training across subsequent sessions was standardized by preferentially increasing speed and then unloading body weight-support. Speed was increased to a range of 2.2 to 2.5 km/h before body weight-support was decreased. There was an active attempt to enhance the level of training at each session. After every Lokomat session, participants performed also 60 minutes of physiotherapy including general exercise program and a conventional gait training
  Interventions: Device: Lokomat (Hocoma, Zurich, Switzerland)
- Control group (Active Comparator): Participants received 25 sessions of conventional physiotherapy. Training occurred approximately 5 days/week for 5 weeks, and each training session lasted 1 hour and half. Patients allocated to the Control Group performed the same conventional physiotherapy training of the other group: a general exercise program and a conventional gait training. The general exercise program consisted in cardiovascular warm-up exercises, muscle stretching exercises, active-assisted or active isometric and isotonic exercises for the main muscles of the trunk and limbs, relaxation exercises, coordination and static/dynamic balance exercises. The conventional gait therapy was based on the proprioceptive neuromuscular facilitation concept, training in walking on different surfaces with or without appropriate walking aids, exercises for the restoration of a correct gait pattern, implementation of residual compensatory strategies and progressive increase of walking resistance
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Device: Lokomat (Hocoma, Zurich, Switzerland) — Patients allocated to the Experimental group performed a Robotic Assisted Gait Training by means of the Lokomat. The Lokomat is robotic device set up as an exoskeleton on the lower limbs of the patient. The system uses a dynamic body weight-support system to support he participant above a motorized treadmill synchronized with the Lokomat.
  Arms: Experimental group
Other: Conventional Physiotherapy — Patients allocated to the Control Group performed a general exercise program and a conventional gait training. The same trained therapist treated all the patients in this group and standardized the duration of each part of the treatment.
  Arms: Control group

SUMMARY:
In Multiple Sclerosis (MS) gait disorders represent one of the most disabling aspect that strongly influence patient quality of life. The improvement of walking ability is a primary goal for rehabilitation treatment. Current promising rehabilitative approaches for neurological disorders are based on the concept of the task-specific repetitive training. Hence, the interest in automated robotic devices that allow this typology of treatment for gait training. However, studies on the effectiveness of such methodologies are still poorly numerous in terms of functional improvement in MS patients. The aim of this controlled cross-over study is to evaluate the effectiveness of a Lokomat gait training in patients affected by Multiple Sclerosis in comparison to a ground conventional gait training.

DETAILED DESCRIPTION:
In Multiple Sclerosis (MS), the highly variable distribution of demyelinization areas and axonal loss in the Central Nervous System can lead to very complex and unpredictable neurological deficits and clinical patterns. Gait disorders as reduced speed and stride length, gait asymmetry, increased muscular energy expenditure, balance deficit and increased risk of falling, represent one of the most disabling aspect. These motor problems strongly influence the level of independence that a person affected by MS is able to achieve, resulting in severe negative impact on quality of life. Therefore, the improvement of walking ability is a primary goal for rehabilitation treatment. Many studies demonstrated that a conventional rehabilitation treatment based on physiotherapy could be effective in increasing muscle strength and motor function, improving gait and mobility abilities, reducing fatigue and risk of falls, leading finally to an overall increase of patient autonomy. According to the most recent neurophysiological concepts based on neural plasticity, in recent years the rehabilitative approaches that seem to be more effective in improving functional performance are based on the concept of the task-specific repetitive training. As in the case of the constraint induced movement therapy (CIMT) for upper limb rehabilitation and the body weight support treadmill training (BWSTT) for the lower, the factors that appear to positively affect patient outcome are the intensity, precocity, repeatability, specificity in a training that incorporates high numbers of repetitions of task-oriented practice. Hence, the interest in automated robotic devices for gait training for MS patients has grown. With their consistent, symmetrical lower-limb trajectories, robotic devices provide many of the proprioceptive inputs that may increase cortical activation and stimulation of Central Pattern Generator (CGPs) in order to improve motor function. The use of robot-assisted-gait-training (RAGT) allows: repetition of specific and stereotyped movements in order to acquire a correct and reproducible gait pattern in conditions of balance and symmetry, early start of treatment using the activity with body weight support, safeguard of the patient with reduction of fear of falling, in order to increase the quantity and quality of the performed exercise while minimizing the intervention of a therapist. However, studies on the effectiveness of such methodologies are still poorly numerous in terms of functional improvement in patients with MS. The aim of this controlled cross-over study is to evaluate the effectiveness of a robot-driven gait orthosis (Lokomat - Hocoma, Inc., Zurich, Switzerland) gait training in patients affected by Multiple Sclerosis in comparison to a ground conventional gait training. The improvement in gait pattern, motor ability and autonomy in the functional activities of daily living will be assessed by using validated clinical and functional scales and quantitative instrumental analysis of gait kinematic parameters

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple sclerosis according to the McDonald's Criteria in stable phase of disease for at least 3 months.
* ability to walk 25 foot without assistance
* EDSS score between 3.5 and 7

Exclusion Criteria:

* exacerbations of the disease in the last 3 months
* deficits of somatic sensation involving the legs
* other neurological, orthopedic or cardiovascular co-morbility
* severe posture abnormalities
* severe-moderate cognitive impairment (Mini Mental State ≤ 21)
* body weight greater than 135 kg;
* height more than 200 cm;
* limb-length discrepancy greater than 2 cm;
* presence of skin lesions on the trunk, pelvis and lower limbs that could interfere with the placement of the electrodes and straps anchoring the Lokomat.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Timed 25 Foot Walk (25FW) | 5 weeks
  Assessment of gait performance in terms of speed. First component of the Multiple Sclerosis Functional Composite (MSCF) scale - leg function / ambulation, for the study and measurement of functional outcomes in clinical trials in patients with multiple sclerosis according to the "Task Force on Clinical Outcomes Assessment of the National Multiple Sclerosis Society "- 1994.

SECONDARY OUTCOMES:
Timed 10 meter walking test (TWT) | 5 weeks
  Assessment of gait performance in terms of speed
6 minute walking test (6MWT) | 5 weeks
  Assessment of gait performance in terms of resistance
Tinetti Test (TT) | 5 weeks
  Assessment of balance and gait ability and the falls risk
Functional Ambulation Categories (FAC) | 5 weeks
  Assessment of ambulation ability
Modified Ashworth scale for lower limbs | 5 weeks
  Assessment of lower limbs spasticity
Modified Motricity Index for lower limbs | 5 weeks
  Assessment of lower limbs motor function
Knee extensor strength (KES) | 5 weeks
  Assessment of knee extensor strength by dynamometer measurement
Double Time Support (DST) | 5 weeks
  kinematic parameter corresponding to the duration of the double support phase of gait cycle, calculated as [ms /%]
Step Length Ratio (SLR) | 5 weeks
  kinematic parameter corresponding to gait symmetry, calculated as the ratio between the step length of both legs (shorter step length / longer step length)
Expanded Disability Status Scale (EDSS) | 5 weeks
  Traditionally used disability scale for multiple sclerosis
Functional Independence Measure (FIM) | 5 weeks
  Assessment of daily activities functional autonomy
Quality of Life Index (QL Index - SF36) | 5 weeks
  Measures of health-related quality of life
Numeric Rating Scale (NRS) | 5 weeks
  Assessment of pain

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Bonassi, MD, Study Chair — HABILITA Zingonia; Cristiano Sconza, MD, Principal Investigator — HABILITA Zingonia
Locations (1):
- HABILITA, Zingonia Di Ciserano, Bergamo, Italy

REFERENCES:
- [Result] Schwartz I, Sajin A, Moreh E, Fisher I, Neeb M, Forest A, Vaknin-Dembinsky A, Karusis D, Meiner Z. Robot-assisted gait training in multiple sclerosis patients: a randomized trial. Mult Scler. 2012 Jun;18(6):881-90. doi: 10.1177/1352458511431075. Epub 2011 Dec 6. PMID 22146609
- [Result] Beer S, Aschbacher B, Manoglou D, Gamper E, Kool J, Kesselring J. Robot-assisted gait training in multiple sclerosis: a pilot randomized trial. Mult Scler. 2008 Mar;14(2):231-6. doi: 10.1177/1352458507082358. Epub 2007 Oct 17. PMID 17942510
- [Result] Lo AC, Triche EW. Improving gait in multiple sclerosis using robot-assisted, body weight supported treadmill training. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):661-71. doi: 10.1177/1545968308318473. PMID 18971381
- [Result] Swinnen E, Beckwee D, Pinte D, Meeusen R, Baeyens JP, Kerckhofs E. Treadmill training in multiple sclerosis: can body weight support or robot assistance provide added value? A systematic review. Mult Scler Int. 2012;2012:240274. doi: 10.1155/2012/240274. Epub 2012 May 30. PMID 22701177
- [Result] Vaney C, Gattlen B, Lugon-Moulin V, Meichtry A, Hausammann R, Foinant D, Anchisi-Bellwald AM, Palaci C, Hilfiker R. Robotic-assisted step training (lokomat) not superior to equal intensity of over-ground rehabilitation in patients with multiple sclerosis. Neurorehabil Neural Repair. 2012 Mar-Apr;26(3):212-21. doi: 10.1177/1545968311425923. Epub 2011 Dec 2. PMID 22140197
- [Result] Wier LM, Hatcher MS, Triche EW, Lo AC. Effect of robot-assisted versus conventional body-weight-supported treadmill training on quality of life for people with multiple sclerosis. J Rehabil Res Dev. 2011;48(4):483-92. doi: 10.1682/jrrd.2010.03.0035. PMID 21674396
- [Result] Pilutti LA, Lelli DA, Paulseth JE, Crome M, Jiang S, Rathbone MP, Hicks AL. Effects of 12 weeks of supported treadmill training on functional ability and quality of life in progressive multiple sclerosis: a pilot study. Arch Phys Med Rehabil. 2011 Jan;92(1):31-6. doi: 10.1016/j.apmr.2010.08.027. PMID 21187202
- [Result] Giesser B, Beres-Jones J, Budovitch A, Herlihy E, Harkema S. Locomotor training using body weight support on a treadmill improves mobility in persons with multiple sclerosis: a pilot study. Mult Scler. 2007 Mar;13(2):224-31. doi: 10.1177/1352458506070663. PMID 17450642
- [Result] Eng J. Sample size estimation: how many individuals should be studied? Radiology. 2003 May;227(2):309-13. doi: 10.1148/radiol.2272012051. PMID 12732691